CLINICAL TRIAL: NCT06434272
Title: The Effectiveness of Low-load Blood Flow Restriction Exercise in Patients With an Acute Achilles Tendon Rupture Treated Non-surgically
Brief Title: Blood Flow Restriction Exercise in Patients With an Achilles Tendon Rupture
Acronym: BEAN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other); Aalborg University Hospital (Other); Gødstrup Hospital (Other); Regionshospitalet Horsens (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BEAN (1-10-72-192-23)
Record Dates: First submitted 2024-05-23; First posted 2024-05-30 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Achilles Tendon Rupture
MeSH Terms: interventions — Blood Flow Restriction Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early initiated Blood Flow Restriction Exercise (Experimental): Receives an intervention in adjunct to usual care in weeks 1-12, and continues with usual care in weeks 13-24.
  Interventions: Other: Early exercise with partial Blood Flow Restriction
- Late initiated Blood Flow Restriction Exercise (Experimental): Receives usual care in weeks 1-12, and receives an intervention in adjunct to usual care weeks 13-24.
  Interventions: Other: Late exercise with partial Blood Flow Restriction

INTERVENTIONS:
Other: Early exercise with partial Blood Flow Restriction — The intervention comprises of 12 weeks of blood flow restriction exercise in weeks 1-12 after injury. Three weekly exercise sessions are performed. Six supervised sessions are provided during the 12 weeks.
  Blood flow restriction of 80% of the limb occlusion pressure required to fully restrict the arterial blood flow is employed.
  The intervention comprises three exercises: Seated leg extension, standing knee flexion, and seated heel-rise performed at home as an adjunct to usual care treatment.
  Each exercise is performed in four sets of 30, 15, 15, +1 repetitions, with the fourth set (+1) being as many repetitions as possible.
  Pause in between sets is 30 seconds. Pause in between exercises are 120 seconds.
  In weeks 13-24, patients in this arm follow usual care treatment.
  Other Names: BFR; BFRE; Blood Flow Restriction Exercise; BFR-T; Blood Floow Restriciton Training; LL-BFR; Low Load Blood Flow Restriction
  Arms: Early initiated Blood Flow Restriction Exercise
Other: Late exercise with partial Blood Flow Restriction — The intervention comprises of 12 weeks of blood flow restriction exercise in weeks 13-24 after injury. Three weekly exercise sessions are performed. Six supervised sessions are provided during the 12 weeks.
  Blood flow restriction of 80% of the limb occlusion pressure required to fully restrict the arterial blood flow is employed.
  The intervention comprises three exercises: Leg press in machine, heel-rise in machine, knee flexion in machine performed at training facilities as an adjunct to usual care treatment. If facilities are unavailable, three home-based exercises will be provided.
  Each exercise, regardless of study arm, is performed in four sets of 30, 15, 15, +1 repetitions, with the fourth set (+1) being as many repetitions as possible.
  In weeks 1-12, patients in this arm follow usual care treatment.
  Other Names: BFR; BFRE; Blood Flow Restriction Exercise; BFR-T; Blood Flow Restriction Training; LL-BFR; Low Load Blood Flow Restriction
  Arms: Late initiated Blood Flow Restriction Exercise

SUMMARY:
The goal of this clinical trial is to gain insights into the effects of Blood Flow Restriction Exercise (BFRE) in patients with an acute Achilles tendon Rupture. The main questions it aims to answer are:

Is BFRE an effective adjunct to usual care when compared with only usual care? When is the optimal timing for initiating BFRE: In the early treatment stage or at the later stage after hospital treatment? Participants will receive an intervention comprising 12 weeks of BFRE as an adjunct to usual care.

* Either in the initial 1-12 weeks after Achilles tendon rupture, or
* In the following 13-24 weeks after Achilles tendon rupture

Researchers will compare the two groups at 13 weeks (3 months) to compare BFRE to usual care, and at 25 weeks (6 months) to compare the two time points for initiating BFRE (early vs. late).

DETAILED DESCRIPTION:
This is an assessor-blinded, randomized, controlled multicenter trial with patients allocated 1:1 to one of two parallel groups, with follow-up times at weeks 13 and 25 after allocation.

Patients with an acute Achilles tendon rupture treated non-surgically are eligible for inclusion. All patients will receive a 12-week BFRE program, either in weeks 1-12 or 13-24 post allocation, as an add-on to usual care.

The BFRE program is performed three times weekly on the injured leg at 80% of the limb occlusion pressure required to restrict the arterial blood flow fully.

Outcome measures are assessed at baseline, week 13, and week 25 after allocation. The primary outcome at the week 13 follow-up is the Single-Leg Heel-Raise test which assesses the patient's ability to raise the heel of the injured leg a minimum of 2 cm. The primary outcome at the week 25 follow-up is the Achilles Total Tendon Rupture Score which assesses the patient's self-reported symptoms and physical activity.

During most of the initial trial phase (weeks 1-12), patients are treated at local hospitals, where recruitment, assessment, and randomization occur. Usual care at the hospitals consists of ankle immobilization with a gradual return to weight-bearing in the following weeks. In the latter half of the trial phase (weeks 13-24), patients have transitioned to municipal care, where usual care includes diverse exercises performed at home or training facilities.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 years or older
* have started initial treatment within 72 hours of Achilles tendon rupture
* understand written and spoken Danish

Exclusion Criteria:

* bilateral Achilles tendon rupture
* previous Achilles tendon rupture in either leg
* decreased lower extremity function, caused by conditions other than Achilles tendon rupture
* treated with fluoroquinolones within the last six months
* treated with corticosteroid injection(s) in the area near the Achilles tendon within the last six months.
* diabetes
* previous diagnosed thrombosis
* Known atherosclerosis in the peripheral arteries of the lower limb
* other reasons for exclusion (cognitive deficits, inability to provide informed consent, requiring cast-treatment due to low compliance regarding gradual wedge removal, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 218 (Estimated)
Dates: Start 2025-01-28 (Actual); Primary Completion 2028-01-09 (Estimated); Study Completion 2028-01-09 (Estimated)

PRIMARY OUTCOMES:
Single-leg heel-rise test | Primary outcome at 13 week test. Measured as a secondary outcome at 25 week test.
  Patient's ability to perform a Single-Leg Heel-rise, defined as the ability to raise the heel of the injured leg at least 2 cm while keeping the knee straight. The test is performed with patients standing on a flat surface with the ankle in a neutral position. Patients will be allowed to keep their balance by lightly touching a wall.
Achilles tendon Total Rupture Score (ATRS) | Primary outcome at 25 week test. It is also measured at baseline through recall of the pre-injury condition and at the 13 week test as a secondary outcome.
  The ATRS is a validated patient-reported, injury-specific questionnaire regarding physical activity and symptoms. The ATRS consists of 10 items scored from 0 (major limitations) to 10 (no limitations), resulting in a score between 0 (worst) to 100 (best).

SECONDARY OUTCOMES:
30 seconds unilateral Sit to Stand test | The test will be performed on both legs at 13 week test and 25 test.
  The unilateral 30 second Sit to Stand test (unilateral 30STS) is a clinical test of lower extremity function. The unilateral 30STS tests how many correct repetitions of a sit to stand from a chair, a patient can complete in 30 seconds
Calf circumference | The measurement will be performed on both legs at 13 week test and 25 test.
  The calf circumference is measured in centimeters (cm) on both legs using a tape measure 15 cm below the medial palpable joint line of the knee. Repeated measurements will be made until a consistent measurement is found.
Thigh circumference | The measurement will be performed on both legs at 13 week test and 25 test.
  Thigh circumference is measured in centimeters (cm) on both legs using a tape measure 10 cm proximal to the apex patella. During measurement patients lay supine on an examination table with knees bent in a 90-degree angle.
Achilles tendon elongation (ATRA) | The test will be performed on both legs at 13 week test and 25 test.
  The Achilles tendon length is indirectly measured by the Achilles tendon resting angle (ATRA), measuring the difference in passive dorsiflexion when lying prone with knees in a 90-degree angle.
Single-leg heel-rise height | The test will be performed on both legs at 13 week test and 25 week test.
  Patient's maximum heel-rise height measured in cm. The test is performed with patients standing on a flat surface with the ankle in a neutral position. Patients will be allowed to keep their balance by lightly touching a wall.
Single-leg heel-rise endurance test | The test will be performed on both legs at 25 week test.
  The maximal number of correct single-leg heel-rise repetitions is measured. The test is performed with patients standing on a flat surface with the ankle in a neutral position. Patients will be allowed to keep their balance by lightly touching the wall.
Tampa Scale of Kinesiophobia 13-items (TSK-13) | TSK-13 is measured at baseline, 13 week test, and 25 test.
  The TSK-13 is a 13-item self-reported measure for fear of movement or reinjury, that has previously been used in patients with Achilles tendon rupture.
International Physical Activity Questionnaire-short form (IPAQ-SF) | IPAQ-SF is measured at baseline through recall of pre-injury condition, 13 week test, and 25 week test.
  The IPAQ-SF consists of 7 items on physical activity as time spent performing vigorous and moder-ate activities, the time spent walking, and time spent sitting during the past week. The IPAQ pro-vides an estimate of the total weekly physical activity measured in MET-minutes per week and total minutes spent sitting.
Adverse events | Measured continously, and evaluated at 13 week test and 25 week test.
  The number of adverse events and serious adverse events will be recorded and reported to a Data Safety Monitoring Board. Adverse events are defined as unexpected medical events related to the initial treatment. Serious adverse event are complications requiring further inpatient care, such as re-rupture of the Achilles tendon, non-union of the Achilles tendon, or deep venous thromboembolism and pulmonary embolism. Muscle soreness or mild pain following exercise is expected and not con-sidered an adverse event.

OTHER OUTCOMES:
Patient Acceptable Symptom State (PASS) | Measured at 25 week test.
  Patients are asked on a questionnaire whether they think their current symptom state is satisfactory (yes/no).
Global rating of change | Measured at 13 week test and 25 week test.
  Perceived effect of intervention is rated on a 7-point likert scale from significantly worse to significantly better.
Exercise adherence and progression | Measured continously, and evaluated at 13 week test and 25 week test.
  Patients' adherence with the exercise sessions (completed sessions) and progression during the intervention period will be recorded in self-reported exercise diaries by the patients. Exercise diaries will also be provided to patients in the control group, to monitor usual care exercise.
Demographic data consisting of sex, age, weight, height, BMI, marital status, employment status, alcohol intake, nicotine intake, injury mechanism, and pre-injury ankle pain condition | Measured at baseline.
  Descriptive demographic data.
Limb Occlusion Pressure | Measured at baseline for the Early BFRE-group, and measured at 13 week test for the Late BFRE-group.
  The pressure required to fully occlude arterial inflow to the working limb will be measured. 80% of the total occlusion pressure will be calculated and applied during exercise.
Drop-out rate | Recorded throughout the study-period, and will be evaluated at 13 week test and 25 week test.
  Number of participants who drop out from the trial during the study-period.
Concomitant exercise performed as part of usual care | Measured continuously and evaluated at the 25 week test.
  Exercise diaries detailing what exercises are performed during usual care after hospital treatment.
EuroQol-5 Dimension-5 Levels (EQ-5D-5L) | EQ-5D-5L is measured at baseline, capturing both the recalled pre-injury condition and the current condition, as well as at the 13-week and 25-week tests.
  The EQ-5D-5L is a generic self-reported measure for health-related quality of life consisting of five dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) with five severity levels each. The total score of the descriptive index and EuroQol Visual Analogue Scale (EQ-VAS) ranges from -0.624 (worst) to 1.000 (best) and 0 (worst imaginable health) to 100 (best imaginable health), respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Bentzen, MHSc, Principal Investigator — University of Aarhus; Inger Mechlenburg, DMSc, Study Director — University of Aarhus; Per H. Gundtoft, MD, PhD, Study Director — Aarhus University Hospital; Stian L. Jørgensen, PT, PhD, Study Director — Regionshospitalet Horsens
Locations (1):
- Aarhus University Hospital, Aarhus N, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Anonymised patient-level data will be made available if required by the scientific journal, in which the results of the trial are published. Additionally, researchers presenting a justified cause for receiving the data can obtain it after a data access agreement has been signed.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data will be available after publication of the trial.
Access Criteria: Data access will be reviewed by the author group. Requesters will be required to sign a data access agreement.